CLINICAL TRIAL: NCT02510131
Title: Is Hyacinth Exercise Better Than Kegel's Exercise in Women With Urinary Incontinence?
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Malaya (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PISA
Record Dates: First submitted 2015-07-20; First posted 2015-07-29 (Estimated); Last update posted 2018-05-22 (Actual); Status verified 2018-05

CONDITIONS: Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pelvic floor exercise (Active Comparator): Participants randomized to Kegel's exercises will be asked to contract their pelvic floor muscle for 1-10 seconds, followed by 10 seconds' relaxation.
  Length of duration of exercise is tailored to individual's ability in contracting her pelvic floor muscle.
  Each cycle is equivalent to 1 contraction and 1 relaxation phase. Participants will be asked to perform 3 sessions per day, and to perform their Kegel exercises at home daily.
  1 session of Kegel's exercise is consists of 20 cycles of slow twitch fibre contraction and 30 repetitions of fast twitch fibre for 1 minute.
  Interventions: Behavioral: Exercises
- Hyacinth exercise (Experimental): In this arm participants are also taught Kegel's exercises but will be additionally taught extra steps which mirrored Muslim's praying steps.
  As well as their Kegel's exercises, participants will be asked to perform the extra steps at least 63 minutes per week.
  Participants may choose to perform these at the same time or at a different time from their Kegel's exercises. Participants will be asked to perform 1 cycle (3 minutes and 1 second) for 3 sessions a day for daily.
  Each cycle is consists of repetition of 4 positions: standing upright- 90 degree bow- prostration-sitting.
  Interventions: Behavioral: Exercises

INTERVENTIONS:
Behavioral: Exercises — To compare Hyacinth exercise with Kegel's exercise in improving urinary incontinence

SUMMARY:
To determine whether Hyacinth exercises are more effective than Kegel's exercise at improving pelvic floor weakness among women aged 55 and above with urinary incontinence.

DETAILED DESCRIPTION:
Individuals who admit to have urinary leakage will be examined to determine the nature of their problem and individuals for whom Kegel exercises are likely to be for benefit will be recruited into this study.

One hundred and eighty women who participants who agree to be randomized to Kegel's or Hyacinth exercises will be randomized.

The treatment allocation will be sealed opaque enveloped and stored in a secure location.

Participants will be blinded from the treatment arm, and as much as possible, participants in different arms of the study would be given different appointment dates to avoid contamination.

Exercises will be prescribed by a trained personnel, and flexibility is added to the routine to enable tailoring to individual lifestyles and choices.

ELIGIBILITY:
Inclusion Criteria:

* Woman aged above 55 with urinary incontinence.

Exclusion Criteria:

* Individuals who are unable or unwilling to provide written informed consent.
* Stage 3 and 4 pelvic organ prolapse.
* Individuals who have physical weakness and are unable to do kegel plus exercises.
* Neuropathic injury of pelvic floor muscles.

Min Age: 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2015-08; Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Female pelvic floor questionnaires scoring | 6 months
  to assess woman's urinary incontinence scoring at 0, 2 and 6 months, to look for improvement from baseline to 6 months after exercises

SECONDARY OUTCOMES:
intravaginal biofeedback measurements | 6 months
  to measure the strength of pelvic floor muscle by Femiscan at 0,2 and 6 months, to look for change from baseline to 6 months after exercises

CONTACTS AND LOCATIONS:
Locations (1):
- University Malaya Medical Center, Kuala Lumpur, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Hay-Smith EJC, Starzec-Proserpio M, Moller B, Aldabe D, Cacciari L, Pitangui ACR, Vesentini G, Woodley SJ, Dumoulin C, Frawley HC, Jorge CH, Morin M, Wallace SA, Weatherall M. Comparisons of approaches to pelvic floor muscle training for urinary incontinence in women. Cochrane Database Syst Rev. 2024 Dec 20;12(12):CD009508. doi: 10.1002/14651858.CD009508.pub2. PMID 39704322